CLINICAL TRIAL: NCT05066776
Title: Liquid Biopsy in Combination With PET/CT Versus PET/CT Alone in Diagnosis of Small Lung Nodules
Brief Title: Liquid Biopsy With PET/CT Versus PET/CT Alone in Diagnosis of Small Lung Nodules
Status: Terminated | Type: Observational
Why Stopped: Withdrawal by sponsor
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Rajesh Shah, Director of Interventional Radiology, Palo Alto Veterans Institute for Research
Other Study IDs: SHANEW_0001
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer; Solitary Pulmonary Nodule; Multiple Pulmonary Nodules
Keywords: PET-CT Scan; Liquid Biopsies
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Pulmonary Nodule: Patients at high-risk of lung cancer found to have a pulmonary nodule 6-20 mm in size.

SUMMARY:
The purpose of this study is to determine if a liquid biopsy, a method of detecting cancer from a blood draw, combined with a PET/CT scan, a type of radiological scan, is better at determining whether a lung nodule is cancerous when compared to a PET/CT scan alone. A PET/CT scan is already used for diagnosis of lung nodules, but its efficacy is uncertain in nodules 6-20 mm in size. Therefore, the PET/CT will be evaluated for its diagnostic ability in lesions this size alone and in combination with a liquid biopsy. Secondarily, a machine learning model will be created to see if the combination of the PET/CT imaging data and the liquid biopsy data can predict the presence of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* ECOG performance status of 0,1, or 2
* Newly discovered lung nodule with:

  1. At least one solid lung nodule measuring 6 mm- 20 mm in greatest diameter detected on screening CT
  2. No single lesion larger than 20 mm in greatest diameter when multiple nodules present
  3. High- or intermediate-risk nodules per American College of Chest Physician (ACCP) guidelines
* Able to provide informed consent

Exclusion Criteria:

* Prior cancer of any type for the previous 3 years
* Prior organ, bone marrow, of hematopoietic stem cell transplant
* Contraindication to administration of [18F]FDG
* Inability to undergo a PET/CT scan
* Ongoing infection, either acute or subacute
* Severe COPD or lung disease requiring home oxygen use
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung nodules found via imaging will be selected from the VA Palo Alto Health Care System.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Comparison of liquid biopsy with PET/CT to PET/CT alone for predicting lung cancer | 24 months
  Determine the sensitivity and specificity of liquid biopsy and PET/CT in combination compared with PET/CT alone for predicting lung cancer for lesions 6 mm- 20 mm in size

SECONDARY OUTCOMES:
ctDNA gene panel ability in detecting lung cancer | 24 months
  Determine the sensitivity and specificity of a ctDNA gene panel in detecting lung cancer for lesions 6 mm- 200 mm in size
DNA methylation liquid biopsy ability in detecting lung cancer | 24 months
  Determine the sensitivity and specificity of DNA methylation liquid biopsy in detecting lung cancer for lesions 6 mm- 20 mm in size
Validate ML classifier for predicting lung cancer | 30 months
  Validate a machine learning (ML) classifier for predicting lung cancer using imaging and clinical data.

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Shah, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] MacMahon H, Naidich DP, Goo JM, Lee KS, Leung ANC, Mayo JR, Mehta AC, Ohno Y, Powell CA, Prokop M, Rubin GD, Schaefer-Prokop CM, Travis WD, Van Schil PE, Bankier AA. Guidelines for Management of Incidental Pulmonary Nodules Detected on CT Images: From the Fleischner Society 2017. Radiology. 2017 Jul;284(1):228-243. doi: 10.1148/radiol.2017161659. Epub 2017 Feb 23. PMID 28240562
- [Background] Kinsinger LS, Anderson C, Kim J, Larson M, Chan SH, King HA, Rice KL, Slatore CG, Tanner NT, Pittman K, Monte RJ, McNeil RB, Grubber JM, Kelley MJ, Provenzale D, Datta SK, Sperber NS, Barnes LK, Abbott DH, Sims KJ, Whitley RL, Wu RR, Jackson GL. Implementation of Lung Cancer Screening in the Veterans Health Administration. JAMA Intern Med. 2017 Mar 1;177(3):399-406. doi: 10.1001/jamainternmed.2016.9022. PMID 28135352
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Huo J, Xu Y, Sheu T, Volk RJ, Shih YT. Complication Rates and Downstream Medical Costs Associated With Invasive Diagnostic Procedures for Lung Abnormalities in the Community Setting. JAMA Intern Med. 2019 Mar 1;179(3):324-332. doi: 10.1001/jamainternmed.2018.6277. PMID 30640382
- [Background] National Comprehensive Cancer Network. NCCN Guidelines Lung Cancer Screening Version 1.2020.
- [Background] Li S, Zhao B, Wang X, Yu J, Yan S, Lv C, Yang Y. Overestimated value of (18)F-FDG PET/CT to diagnose pulmonary nodules: Analysis of 298 patients. Clin Radiol. 2014 Aug;69(8):e352-7. doi: 10.1016/j.crad.2014.04.007. Epub 2014 May 27. PMID 24877581
- [Background] Cescon DW, Bratman SV, Chan SM, Siu LL. Circulating tumor DNA and liquid biopsy in oncology. Nat Cancer. 2020 Mar;1(3):276-290. doi: 10.1038/s43018-020-0043-5. Epub 2020 Mar 20. PMID 35122035
- [Background] Nair VS, Keu KV, Luttgen MS, Kolatkar A, Vasanawala M, Kuschner W, Bethel K, Iagaru AH, Hoh C, Shrager JB, Loo BW Jr, Bazhenova L, Nieva J, Gambhir SS, Kuhn P. An observational study of circulating tumor cells and (18)F-FDG PET uptake in patients with treatment-naive non-small cell lung cancer. PLoS One. 2013 Jul 5;8(7):e67733. doi: 10.1371/journal.pone.0067733. Print 2013. PMID 23861795
- [Background] Odahowski CL, Zahnd WE, Eberth JM. Challenges and Opportunities for Lung Cancer Screening in Rural America. J Am Coll Radiol. 2019 Apr;16(4 Pt B):590-595. doi: 10.1016/j.jacr.2019.01.001. PMID 30947892
- [Background] Spalluto LB, Lewis JA, LaBaze S, Sandler KL, Paulson AB, Callaway-Lane C, Grogan EL, Massion PP, Roumie CL. Association of a Lung Screening Program Coordinator With Adherence to Annual CT Lung Screening at a Large Academic Institution. J Am Coll Radiol. 2020 Feb;17(2):208-215. doi: 10.1016/j.jacr.2019.08.010. Epub 2019 Sep 6. PMID 31499025
- [Background] Triplette M, Thayer JH, Pipavath SN, Crothers K. Poor Uptake of Lung Cancer Screening: Opportunities for Improvement. J Am Coll Radiol. 2019 Apr;16(4 Pt A):446-450. doi: 10.1016/j.jacr.2018.12.018. Epub 2019 Feb 15. PMID 30777648
- [Background] Ruilong Z, Daohai X, Li G, Xiaohong W, Chunjie W, Lei T. Diagnostic value of 18F-FDG-PET/CT for the evaluation of solitary pulmonary nodules: a systematic review and meta-analysis. Nucl Med Commun. 2017 Jan;38(1):67-75. doi: 10.1097/MNM.0000000000000605. PMID 27741214
- [Background] Tang K, Wang L, Lin J, Zheng X, Wu Y. The value of 18F-FDG PET/CT in the diagnosis of different size of solitary pulmonary nodules. Medicine (Baltimore). 2019 Mar;98(11):e14813. doi: 10.1097/MD.0000000000014813. PMID 30882661
- [Background] Constancio V, Nunes SP, Henrique R, Jeronimo C. DNA Methylation-Based Testing in Liquid Biopsies as Detection and Prognostic Biomarkers for the Four Major Cancer Types. Cells. 2020 Mar 5;9(3):624. doi: 10.3390/cells9030624. PMID 32150897